CLINICAL TRIAL: NCT05732285
Title: A Pilot Randomized Controlled Trial of A Comprehensive Cognitive and Affective Intervention for Neurocognitive Disorders (CoINTEGRATE)
Brief Title: A Pilot Randomized Controlled Trial: CoINTEGRATE
Acronym: CoINTEGRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hala Darwish, Associate Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00210257
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Neurocognitive Disorders; Cognitive Dysfunction; Traumatic Brain Injury; Multiple Sclerosis; Mild Cognitive Impairment
Keywords: Affective Dysfunction; Cognitive Behavioral Therapy; Modifiable lifestyle factors; Cognitive Rehabilitation Therapy; Long COVID (coronavirus disease)
MeSH Terms: conditions — Neurocognitive Disorders; Cognitive Dysfunction; Brain Injuries, Traumatic; Multiple Sclerosis; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: CRT plus CBT plus lifestyle modification or usual care
Who Masked: Care Provider
Masking Description: Only the data collectors in this study will be blind to the patient's group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CRT plus CBT and Lifestyle modifications (Experimental)
  Interventions: Behavioral: CRT; Behavioral: CBT; Behavioral: Modifiable lifestyle factors
- Usual care (Active Comparator)
  Interventions: Behavioral: Usual care Psychoeducation

INTERVENTIONS:
Behavioral: CRT — Participants that score 1-1.5 standard deviation (SD) below the norm for age and education on 2 cognitive domains will receive an intensive program, 2 CRT sessions per week for 4 weeks in addition to 1 CBT session per week for 8 weeks. Based on clinical experience, those with more severe cognitive deficits require more time to achieve their therapy goals, whereas those with mild deficits can tolerate a more intense therapy.
  Participants that score 1.5-2 SD or more below the norm for age and education on 2 cognitive domains will receive 1 CRT and 1 CBT weekly sessions for 8 weeks. All the CRT sessions will be coupled with homework for 8 weeks.
  All research-related sessions will be web-based (on Zoom) and recorded (with approval).
  Arms: CRT plus CBT and Lifestyle modifications
Behavioral: CBT — Participants that score 1-1.5 standard deviation (SD) below the norm for age and education on 2 cognitive domains will receive an intensive program, 2 CRT sessions per week for 4 weeks in addition to 1 CBT session per week for 8 weeks. Based on clinical experience, those with more severe cognitive deficits require more time to achieve their therapy goals, whereas those with mild deficits can tolerate a more intense therapy.
  Participants that score 1.5-2 SD or more below the norm for age and education on 2 cognitive domains will receive 1 CRT and 1 CBT weekly sessions for 8 weeks. All the CRT sessions will be coupled with homework for 8 weeks.
  All research-related sessions will be web-based (on Zoom) and recorded (with approval).
  Arms: CRT plus CBT and Lifestyle modifications
Behavioral: Modifiable lifestyle factors — The therapy sessions are coupled with homework and requires some lifestyle modifications such lifestyle adjustments are using a calendar, a diary, maintaining a sleep schedule and exercise.
  Arms: CRT plus CBT and Lifestyle modifications
Behavioral: Usual care Psychoeducation — Participants will receive 15 minute psychoeducation session twice per week for 8 weeks.
  All research-related sessions will be web-based (on Zoom) and recorded (with approval).
  Arms: Usual care

SUMMARY:
The purpose of this study is to examine the feasibility of comprehensive multimodal individually tailored Cognitive Behavioral Therapy (CBT), Cognitive Rehabilitation Therapy (CRT), and modifiable lifestyle sessions.

The study team hypothesizes that combining evidence-based cognitive and affective therapies with lifestyle modifications is feasible and will improve the community integration (CI) and Quality of life (QoL) in patients with a neurocognitive disorder compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with one of the following: Mild Trauma Brain injury (TBI), Multiple Sclerosis (MS), Long COVID, or Mild Cognitive Impairment (MCI)
* MCI patients age older than 50 years old, all other diagnosis 21-65 years old and are receiving care through the Michigan medicine network
* Participants that can provide consent or legally authorized representative who can provide consent on their behalf
* Cognitive impairment ≥ 1.0 standard deviation below the test score normed for age and education in at least 2 cognitive domains (verbal learning and memory, processing speed, or visuospatial memory)

Exclusion Criteria:

* TBI participants symptomatic at rest (headache, dizziness, nausea, or vertigo) will be referred to primary care physician (PCP)
* History of TBI (except for participants with TBI)
* MS participants with recent relapse (1 month prior to enrollment) or on Intravenous or oral steroids
* MCI participants with disease duration greater than 1 year
* Patients with other neurosensory or neurodegenerative diseases
* Diagnosed with COVID-19 (except for Long COVID group)
* Psychiatric disorders other than mild to moderate anxiety and depression
* Patients with severe depression or suicidal (ideation or plan) will be instructed to seek mental health, provided with resources and referred to patient's primary care provider
* Diagnosed sleep disorders
* Visual or auditory impairment,
* Current or history of alcohol or substance abuse/dependence
* Cognitive impairment less than 1.0 standard deviation below the test score normed for age and education in at least 2 cognitive domains (verbal learning and memory, processing speed, or visuospatial memory)
* Cognitive impairment greater or equal to 1.0 standard deviation below the test score normed for age and education in 1 cognitive domain (verbal learning and memory, processing speed, or visuospatial memory)
* Currently receiving CRT, CBT or Occupational therapy (OT) or another type of psychological therapy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Number of patients that complete the study | week 8 (end of treatment)
Average number of sessions completed | week 8 (end of treatment)
Overall experience based qualitative semi-structured interview | Week 9 (after treatment ended)
  This interview will be conducted at the end of the study and in the order of exit of participants to gather feedback about their satisfaction with the study. This brief interview consists of 3 questions that ask the participants to describe the aspects of the intervention participants found beneficial, willingness to participate again, and whether it was appropriate for participants needs. In addition, a brief quantitative satisfaction survey to rate overall satisfaction, how likely it would be recommend to others, and how satisfied participants are with telemedicine as a mode of delivery.

SECONDARY OUTCOMES:
The Community Integration Questionnaire (CIQ) Score | Week 9 (after treatment ended)
  This questionnaire contains 15 items to evaluate the degree of integration into each of the three area of home, social network, and productive activities. The overall score, which represents a summation of the home integration score plus social integration score plus productivity score, can range from 0 to 29. A high score indicates greater integration, and a low score reflects less integration.
The Short Form Health Survey (SF-36) | Week 9 (after treatment ended)
  The SF-36 explores people's physical and mental health. It consists of 36 items that assess role limitations due to personal or emotional problems, emotional well-being, social functioning, general health perceptions, perceived change in health. Scores ranged from 0 (worst health status) to 100 (best health status).
Montreal Cognitive Assessment (MoCA) | Week 9 (after treatment ended)
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
The Symbol Digit Modalities Test Score (SDMT-5 minutes) | Week 9 (after treatment ended)
  The Symbol Digit Modalities Test (SDMT) is used to assess divided attention, visual scanning, tracking and motor speed. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Because examinees can give either written or spoken responses, the test is well suited for use with individuals who have motor disabilities or speech disorders. Because it involves only geometric figures and numbers, the SDMT is relatively culture free as well and can be administered to individuals who do not speak English. It takes approximately 5 minutes to complete the entire test. Scoring involves summing the number of correct substitutions within the 90 second interval the max score is 110, where a higher score indicates a better memory.
Brief Visuospatial Memory test (BVMT-R-25 minutes) | Week 9 (after treatment ended)
  This test is comprised of three memory trials (10 seconds each) followed by delayed recall after 25 minutes and a recognition trial. It has been widely used as a quick measure of visuospatial memory. The digital stimulus forms will be used (alternate form will be used at the end of the study to control for practice effect).
  Recall performance will record for each of the immediate recall trials (Trial 1, Trial 2, and Trial 3) and for the delayed recall trial (Delayed Recall). The study team will combine the recall scores to form three additional summary measures of learning and memory. Recognition Hits and False Alarms will be recorded during the delayed recognition task. Recognition Hits are calculated as the number of correct responses to target items, and Recognition False Alarms are calculated as the number of incorrect responses to nontarget items. Each trial is worth 0-12 points, so the total score is 0-36, a higher score indicates a better memory.
California Verbal Learning Test-Third Edition (CVLT-3-60 minutes) | Week 9 (after treatment ended)
  The California Verbal Learning Test, Third Edition (CVLT-3) measures both recall and recognition of two lists of words (List A and List B) over a number of immediate and delayed memory trials. It provides an assessment of verbal learning and memory deficits in adults ages 16 - 90. Score of 0-16, where a lower score indicates worse memory, and a high score indicates better memory.
The Memory Complaint Scale (MCS-2 minute) score | Week 9 (after treatment ended)
  The Memory Complaint Scale (MCS-2 min) is comprised of 14 items and is designed for subjective memory complaints.The test yields a total score with a classification in terms of memory complaint (MC) based on their score as follows: No MC (0-2), mild MC (3-6), moderate MC (7-10) or severe MC (11-14).

CONTACTS AND LOCATIONS:
Overall Officials: Hala Darwish, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No